CLINICAL TRIAL: NCT06082401
Title: Evaluating the Addition of Hemodiafiltration to Ex-vivo Lung Perfusion - Impact on the Regeneration of Marginal Donor Lungs: a Prospective Randomized Pilot Study
Brief Title: Evaluating the Addition of Hemodiafiltration to EVLP - Impact on the Regeneration of Marginal Donor Lungs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: XVIVO Perfusion (Industry)
Responsible Party: Principal Investigator, Alberto Benazzo, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FILONEX
Record Dates: First submitted 2023-01-04; First posted 2023-10-13 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Hemodiafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): EVLP + HDF
  Interventions: Device: hemodiafiltration (HDF); Device: Ex vivo lung perfusion (EVLP)
- Control Group (Active Comparator): EVLP
  Interventions: Device: Ex vivo lung perfusion (EVLP)

INTERVENTIONS:
Device: hemodiafiltration (HDF) — Hemodiafiltration (HDF) is a variation of conventional HD. By the addition of a substitution solution, convection forces are significantly increased. This substitution solution is added to the blood and is completely removed again in the dialyzer. This increases the negative pressure on the dialysate side and the removal of toxins through convection. The substitution solution can be added in a pre-dilution (before the dialyzer) or post-dilution (after the dialyzer) manner. Pre-dilution is associated with longer run times, less filter clotting, but is also less effective in removing toxins. Post-dilution offers a better toxin clearance capacity, but is associated with an increased risk of filter clotting. Several studies have shown that HDF provides higher clearance rates for both small and middle molecule solutes. Moreover, effective cytokine removal has been shown in HDF both in acute and chronic renal disease patients.
  Other Names: device: multiFiltrate Ci-Ca(R) (by Fresenius)
  Arms: Treatment Group
Device: Ex vivo lung perfusion (EVLP) — Lung transplantation has become a standard treatment for patients suffering from end-stage lung diseases. One of the major obstacles in the modern transplant era is the fact that the need for organs by far exceeds availability. This leads to growing waiting lists with mortality rates ranging between 10-30%. On the other hand, up to 80% of offered lungs from brain dead donors are rejected because they do not meet predefined donor selection criteria.
  Recently, ex vivo lung perfusion (EVLP) has become available as a tool to expand the donor pool. Based on experimental work by Stig Steen, the Toronto lung transplant group developed an EVLP system with the purpose to evaluate lungs with uncertain quality. Consequently, Aigner et al. have expanded the indications for EVLP by showing that primarily unacceptable donor lungs can be reconditioned and then become suitable for transplantation. This concept of organ repair by EVLP has recently been highlighted by a number of publications.
  Other Names: device: XPS (TM) (by XVIVO)

SUMMARY:
The primary objective of the study is the evaluation of the effect of hemodiafiltration during ex vivo lung perfusion in marginal donor lungs, and its feasibility. The hypothesis of this study is that this therapy could stabilize perfusate electrolyte composition, remove toxins and waste products, normalize pH levels and prevent edema formation, thereby reconditioning marginal donor lungs for transplantation.

The proposed pilot study addresses the unmet clinical needs in several aspects: a) for the first time a homeostatic device will be introduced in EVLP to reach stable perfusate composition; b) the proposed modification of the standard EVLP could lead to longer perfusion times, making elective transplantation possible and setting the base for possible ex vivo lung treatments; c) the ultimate effect of the proposed study is to increase organ availability through reconditioning of marginal donor lungs.

ELIGIBILITY:
Inclusion Criteria:

* Marginal donor lungs according to the ISHLT criteria (18)

  * PaO2/FiO2 ratio < 400 (with FiO2=1.0 and PEEP=5-8cmH2O)
  * Donor age ≥ 55 years
  * Smoking history ≥ 20 pack-years
  * Infiltrates in chest radiograph
  * Significant secretions in bronchoscopy
  * Organisms on sputum gram stain
* Donor age > 18 years

Exclusion Criteria:

For donor organs:

* Bilateral consolidations in donor lungs
* Lungs from donors with chest trauma
* Lungs from drowned donors

For patients receiving lung transplantation:

* Inclusions in other interventional studies
* Patients on the intensive care unit (ICU) prior to transplantation, with mechanical ventilation and/or extracorporeal membrane oxygenation (ECMO) support
* Re-transplantations

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
suitability for transplantation of the lungs after 6 hours of EVLP with HDF | 6 hours
PGD grade 3 at 72 hours after transplantation | 72 hours
  for all transplanted organs

SECONDARY OUTCOMES:
survival | months
  survival assessed at 12 and 24 months
Length of mechanical ventilation | up to 100 days
length of ICU stay | up to 100 days
length of hospital stay | up to 200 days
lung function parameters (MEF50) | 24 months
  1, 3, 6, 12 and 24 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Benazzo, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No